CLINICAL TRIAL: NCT01943058
Title: A Phase II Head-to-Head Comparison of Fertility-Sparing Approaches to Treat Complex Atypical Hyperplasia of the Edometrium: Megestrol Versus Levonorgestrel-Releasing Intrauterine System (LNG-IUS)
Brief Title: Megestrol Acetate or Levonorgestrel-Releasing Intrauterine System in Treating Patients With Atypical Endometrial Hyperplasia or Endometrial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5U-12-1; NCI-2013-01725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 5U-12-1 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Atypical Endometrial Hyperplasia; Endometrial Adenocarcinoma; Recurrent Endometrial Carcinoma; Stage IA Endometrial Carcinoma; Stage IB Endometrial Carcinoma; Stage II Endometrial Carcinoma; Stage IIIA Endometrial Carcinoma; Stage IIIB Endometrial Carcinoma; Stage IIIC Endometrial Carcinoma; Stage IVA Endometrial Carcinoma; Stage IVB Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (megestrol acetate) (Experimental): Patients receive megestrol acetate PO BID for up to 18 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: megestrol acetate; Other: laboratory biomarker analysis; Other: questionnaire administration
- Arm B (levonorgestrel-releasing IUS) (Experimental): Patients receive levonorgestrel-releasing IUS with continuous release for up to 18 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Device: levonorgestrel-releasing intrauterine system; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Drug: megestrol acetate — Given PO
  Other Names: BDH 1298; Maygace; Megace; Megestil; Niagestin
  Arms: Arm A (megestrol acetate)
Device: levonorgestrel-releasing intrauterine system — Given IUD
  Other Names: Mirena
  Arms: Arm B (levonorgestrel-releasing IUS)
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well megestrol acetate or levonorgestrel-releasing intrauterine system works in treating patients with atypical endometrial hyperplasia or endometrial cancer. Progesterone can cause the growth of endometrial cancer cells. Hormone therapy using megestrol acetate or levonorgestrel-releasing intrauterine system may fight endometrial cancer by lowering the amount of progesterone the body makes. It is not yet known whether megestrol acetate is more effective than levonorgestrel-releasing intrauterine system in treating atypical endometrial hyperplasia or endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the levonorgestrel-releasing intrauterine system (IUS) results in histologic regression of the endometrial lesion (complex atypical hyperplasia [CAH] and grade 1 endometrial cancer [EC]) comparable to that achieved with oral megestrol (megestrol acetate).

SECONDARY OBJECTIVES:

I. To compare both the side effect profiles, such as weight gain and mood changes as well as compliance with assigned treatment between the 2 treatment arms.

TERTIARY OBJECTIVES:

I. To describe fertility-related outcomes, ovulation, menstrual pattern and fertility abnormalities determined during usual workup (e.g., semen analysis), pregnancy and delivery within 18-months of treatment.

II. To characterize the incidence of endocrine comorbidities (e.g., hypothyroidism, polycystic ovarian syndrome, and diabetes).

III. To characterize the association of levels of endoplasmic reticular (ER) stress and protein kinase B (Akt)-activation in endometrial samples with clinicopathologic-response to Progestin (therapeutic progesterone) therapy.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive megestrol acetate orally (PO) twice daily (BID) for up to 18 months in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive levonorgestrel-releasing IUS with continuous release for up to 18 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of complex atypical hyperplasia or grade 1 endometrioid adenocarcinoma of the endometrium diagnoses within 3 months of study enrollment who strongly desire to maintain fertility
* A diagnosis of endometrioid adenocarcinoma will undergo a magnetic resonance imaging (MRI) scan of the pelvis to rule out deep (> 50%) myometrial invasion and extrauterine metastases
* A negative urine or serum pregnancy test at the time of enrollment
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; a female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Willing and able to consent for treatment with office endometrial biopsies every 3 months
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* A diagnosis of grade 1 endometrioid adenocarcinoma of the endometrium who does not wish to maintain fertility
* MRI evidence of deep myometrial and/or extrauterine spread
* Congenital or other structural uterine or tubal abnormality
* An acute pelvic inflammatory disease or medical conditions, such as, but not limited to acquired immunodeficiency syndrome (AIDS) and chronic immunosuppression, that may be associated with an increased susceptibility to infections
* Current diagnosis of breast cancer or any other cancer
* Currently pregnant or breastfeeding
* Thromboembolic disease, deep vein thrombosis, hypercoagulable state

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Histologic regression from endometrioid adenocarcinoma or complex atypical hyperplasia to benign endometrium | Up to 6 months after completion of study treatment
  Histologic regression will be dichotomized as a binary outcome variable, yes if patients have a confirmed histologic regression at the time of the scheduled biopsy, and no if the histologic regression is not observed regardless of compliance, lost-to-follow-up, or other issues. A contingency table and a bar plot will be used to show the histologic regression rate between the 2 arms. Two-group test of equivalence in proportions will be used to detect whether the histologic regression rate in Arm B is not significantly lower than that in Arm A.

SECONDARY OUTCOMES:
Change in weight | Baseline to up to 6 months after completion of study treatment
  Weight gain will be recorded longitudinally at each 3-month clinic visit and body mass index (BMI) will be calculated and analyzed over time. Can be evaluated using chi squared tests, logistic regression, or repeated measures analysis of variance (ANOVA) whenever appropriate.
Change in mood ascertained using the self-reported Beck Depression Inventory-Primary Care (BDI-PC) | Baseline to up to 6 months after completion of study treatment
  Can be evaluated using chi squared tests, logistic regression, or repeated measures ANOVA whenever appropriate.
Compliance | Up to 6 months after completion of study treatment
  Can be evaluated using chi squared tests, logistic regression, or repeated measures ANOVA whenever appropriate.

OTHER OUTCOMES:
Change in levels of ER stress | Baseline up to 6 months after completion of study treatment
  The changes in the biomarker levels will be examined using scatter plots or tables and paired tests such McNemar test, paired t-test or repeated measures ANOVA whenever appropriate.
Changes in levels of tumorigenic biomarkers | Baseline up to 6 months after completion of study treatment
  The changes in the biomarker levels will be examined using scatter plots or tables and paired tests such McNemar test, paired t-test or repeated measures ANOVA whenever appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lin-Liu, Principal Investigator — University of Southern California